CLINICAL TRIAL: NCT07034430
Title: Genetic Risk Stratification in Ascending Aortic Dilatation Below Surgical Threshold: A Retrospective Single-Center Study
Brief Title: Aortic Dilatation Under 5 cm: Genetic Risk Mapping
Status: Active, not recruiting | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: GOKAEK-2025/9/2
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Ascending Aortic Dilatation; Aortic Aneurysm, Thoracic; Aortic Diseases
Keywords: Non-Syndromic Aortopathy; Syndromic Aortopathy; Aortic Root Dilatation; Next Generation Sequencing (NGS); Borderline Aortic Diameter
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aortic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples will be retained for DNA extraction. Genomic DNA isolated from these samples will be used for targeted analysis of syndromic and non-syndromic aortopathy gene panels using Next Generation Sequencing (NGS). All biospecimens will be stored at -80°C and may be used for future genetic analysis related to aortic disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aortic Dilatation Group: Patients with ascending aortic diameter between 4.0-5.0 cm Retrospectively analyzed for syndromic and non-syndromic genetic mutations using NGS
- Control Group: Population-based exome data from individuals without aortic disease Used for comparison of variant frequency and mutation prevalence

SUMMARY:
This retrospective study investigates the prevalence of genetic mutations in patients with ascending aortic dilatation measuring between 4.0 and 5.0 cm-below the standard surgical threshold. Using Next Generation Sequencing (NGS), both syndromic and non-syndromic aortopathy gene panels were analyzed in 102 patients who had no history of aortic surgery, dissection, or known genetic disorders. Findings will be compared with population data to better understand genetic risk profiles in borderline aortic dilatation, potentially supporting earlier interventions based on genetic markers. The study was approved by the Samsun University Non-Interventional Clinical Research Ethics Committee (GOKAEK, 2025/9/2).

DETAILED DESCRIPTION:
This retrospective study aims to investigate the prevalence of syndromic and non-syndromic genetic mutations in patients with borderline ascending aortic dilatation (aortic diameter between 4.0-5.0 cm). The study cohort includes patients evaluated at Samsun Training and Research Hospital between 2020 and 2025 who underwent genetic testing using targeted Next Generation Sequencing (NGS) panels for aortopathy. The inclusion criteria focus on individuals aged 20-70 years without known connective tissue syndromes or aortic surgery history. The goal is to identify pathogenic or likely pathogenic variants in known aortopathy-associated genes and correlate these findings with patient-specific factors such as age, sex, and aortic measurements.The outcomes of this study may contribute to earlier identification and stratification of genetic risk in patients with aortic dilation below current surgical thresholds, potentially guiding future recommendations for genetic screening and elective surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-70 years
* Ascending aortic diameter between 4.0-5.0 cm
* Underwent genetic panel testing
* No prior aortic surgery
* No history of dissection or rupture
* No known vasculitis or genetic syndrome

Exclusion Criteria:

* Age <20 or >70
* Emergency surgical indication
* Active infection or metabolic instability
* No available genetic test results

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients aged 20 to 70 years who were evaluated at the Samsun Training and Research Hospital's Cardiovascular Surgery, Cardiology, or Medical Genetics outpatient clinics between 2020 and 2025. All patients have an ascending aortic diameter between 4.0 and 5.0 cm on echocardiography or thoracoabdominal CT imaging and underwent genetic testing for syndromic or non-syndromic aortopathy panels. Patients with prior aortic surgery, known genetic syndromes, acute aortic events (rupture or dissection), or vasculitis were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of Syndromic and Non-Syndromic Genetic Mutations | 12 months (Proportion of patients with identified mutations from the genetic panel using NGS.)
  Assessment of the prevalence of genetic mutations associated with syndromic and non-syndromic aortopathies among patients with ascending aortic diameters between 4.0 and 5.0 cm.

SECONDARY OUTCOMES:
Correlation Between Specific Genetic Mutations and Aortic Diameter | 12 months (Statistical correlation coefficients and p-values for associations between variants and patient characteristics.)
  To assess whether certain mutations are associated with larger aortic diameters within the 4.0-5.0 cm range. Evaluation of associations between specific genetic variants and clinical variables such as age, sex, body mass index, and ascending aortic diameter.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Sezer, Principal Investigator — Samsun University Faculty of medicine
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)